CLINICAL TRIAL: NCT02648087
Title: Prevalence of Sleep-disordered Breathing in Patients With a Newly Diagnosed Non Small Cell Lung Cancer
Acronym: NEOSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015 -A00395 - 44
Record Dates: First submitted 2015-11-27; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Bronchial Cancer
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- With and without SDB (Other): comparison of patients with and without sleep-disordered breathing
  Interventions: Device: With and without SDB

INTERVENTIONS:
Device: With and without SDB — Screening of sleep-disordered breathing (SDB)

SUMMARY:
There is a possible implication of sleep apnea syndrome via night-time intermittent hypoxemia in perturbation of quality of life and tumour progression to patients with a bronchial cancer.

The aim of the study is to evaluate this possibility with the help of a night record of sleep and quality of life questionnaires.

DETAILED DESCRIPTION:
There is a possible implication of sleep apnea syndrome via night-time intermittent hypoxemia in perturbation of quality of life and tumour progression to patients with a bronchial cancer.

Enrollment 1200 patients This wide sample is expected to respond to the main and secondary objectives of the study

ELIGIBILITY:
Inclusion Criteria:

* patients with NSCLC undergoing diagnostic
* Performance status 0,1,2

Exclusion Criteria:

* >75 years
* OSA known and in the last 12 months treated PS >2
* Patients under a long-term oxygen therapy
* persons deprived of liberty by judicial decision.
* <18 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation index | Between day 1 and day 15
  RECORDING BY POLYGRAPHY DEVICE between day 1 and day 15 after enrollment